CLINICAL TRIAL: NCT05304585
Title: A Prospective Phase 3 Study of Patients With Newly Diagnosed Very Low-Risk and Low-Risk Fusion Negative Rhabdomyosarcoma
Brief Title: Chemotherapy for the Treatment of Patients With Newly Diagnosed Very Low-Risk and Low Risk Fusion Negative Rhabdomyosarcoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARST2032; NCI-2022-01012 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ARST2032 (Other: Children's Oncology Group); ARST2032 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2022-02-24; First posted 2022-03-31 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-10

CONDITIONS: Embryonal Rhabdomyosarcoma; Fusion-Negative Alveolar Rhabdomyosarcoma; Spindle Cell/Sclerosing Rhabdomyosarcoma
MeSH Terms: conditions — Rhabdomyosarcoma, Embryonal | interventions — Biopsy; Cyclophosphamide; Dactinomycin; Magnetic Resonance Spectroscopy; Radiotherapy; Radiation; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Regimen M (positive mutation) (Experimental): Patients receive vincristine IV on day 1 of each cycle and days 8 and 15 of cycles 2-4, 7-8, and 11-12 and dactinomycin IV over 1-5 minutes or 10-15 minutes on day 1 of cycles 2-5 and 8-14. Patients also receive cyclophosphamide IV over 60 minutes on day 1 of each cycle. Treatment repeats every 21 days for 12-13 cycles in the absence of disease progression or unacceptable toxicity. Patients may also undergo radiation therapy at cycle 5. Patients undergo CT scan, MRI, bone scan, PET scan and tumor biopsy throughout the study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Bone Scan; Procedure: Computed Tomography; Drug: Cyclophosphamide; Biological: Dactinomycin; Procedure: Magnetic Resonance Elastography; Procedure: Positron Emission Tomography; Radiation: Radiation Therapy; Drug: Vincristine
- Regimen VA (VLR RMS) (Experimental): Patients with VLR RMS receive vincristine intravenously (IV) on day 1 of each cycle and days 8 and 15 of cycles 1, 3, 5, and 7 and dactinomycin IV over 1-5 minutes or over 10-15 minutes on day 1 of each cycle. Treatment repeats every 21 days for 8 cycles in the absence of disease progression or unacceptable toxicity. Patients with MYOD1 or TP53 mutated tumors transition to Regimen M at cycle 2 (if mutation status is determined to be positive at week 3) or cycle 3 (if mutation status is determined to be positive after week 3). Patients undergo CT scan, MRI, bone scan, PET scan and tumor biopsy throughout the study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Bone Scan; Biological: Dactinomycin; Procedure: Magnetic Resonance Elastography; Procedure: Positron Emission Tomography; Drug: Vincristine
- Regimen VAC/VA (VL RMS) (Experimental): Patients with LR RMS receive vincristine IV on day 1 of each cycle and days 8 and 15 of cycles 1-3. Patients also receive dactinomycin IV over 1-5 minutes or 10-15 minutes and cyclophosphamide IV over 60 minutes on day 1 of each cycle. Treatment repeats every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive vincristine IV on day 1 of each cycle and days 8 and 15 of cycles 5-7 and dactinomycin IV over 1-5 minutes or over 10-15 minutes on day 1 of each cycle. Treatment repeats every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients with MYOD1 or TP53 mutated tumors transition to Regimen M at cycle 2 (if mutation status is determined to be positive at week 3) or cycle 3 (if mutation status is determined to be positive after week 3). Radiation therapy (if needed) will be administered at cycle 5.Patients undergo CT scan, MRI, bone scan, PET scan and tumor biopsy throughout the study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Bone Scan; Procedure: Computed Tomography; Drug: Cyclophosphamide; Biological: Dactinomycin; Procedure: Magnetic Resonance Elastography; Procedure: Positron Emission Tomography; Drug: Vincristine

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo tumor biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
  Arms: Regimen M (positive mutation); Regimen VAC/VA (VL RMS)
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
  Arms: Regimen M (positive mutation); Regimen VAC/VA (VL RMS)
Biological: Dactinomycin — Given IV
  Other Names: Actinomycin A IV; Actinomycin C1; Actinomycin D; Actinomycin I1; Actinomycin IV; Actinomycin X 1; Actinomycin-[thr-val-pro-sar-meval]; Cosmegen; DACT; Dactinomycine; Lyovac Cosmegen; Meractinomycin
Procedure: Magnetic Resonance Elastography — Undergo MRI
  Other Names: MRE
Procedure: Positron Emission Tomography — Undergo PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Radiation: Radiation Therapy — Undergo radiation
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
  Arms: Regimen M (positive mutation)
Drug: Vincristine — Given IV
  Other Names: LCR; Leurocristine; VCR; Vincrystine

SUMMARY:
Rhabdomyosarcoma is a type of cancer that occurs in the soft tissues in the body. This phase III trial aims to maintain excellent outcomes in patients with very low risk rhabdomyosarcoma (VLR-RMS) while decreasing the burden of therapy using treatment with 24 weeks of vincristine and dactinomycin (VA) and examines the use of centralized molecular risk stratification in the treatment of rhabdomyosarcoma. Another aim of the study it to find out how well patients with low risk rhabdomyosarcoma (LR-RMS) respond to standard chemotherapy when patients with VLR-RMS and patients who have rhabdomyosarcoma with DNA mutations get separate treatment. Finally, this study examines the effect of therapy intensification in patients who have RMS cancer with DNA mutations to see if their outcomes can be improved.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the failure free survival (FFS) of patients with very low-risk (VLR) rhabdomyosarcoma (RMS) (fusion negative [FN], stage 1, clinical group [CG] I, MYOD1 wildtype [WT], TP53 [WT]) when treated with 24 weeks of vincristine and dactinomycin (VA).

II. To evaluate the FFS of patients with low-risk (LR) RMS (FN, stage 1 CG II, or stage 2 CG I/II or CG III [orbit only], MYOD1 WT, TP53 WT) when treated with 12 weeks of vincristine, dactinomycin and cyclophosphamide (VAC) followed by 12 weeks of VA.

SECONDARY OBJECTIVES:

I. To evaluate the overall survival (OS) of patients with VLR RMS treated with 24 weeks of VA.

II. To evaluate the OS of patients with LR RMS treated with 12 weeks of VAC followed by 12 weeks of VA.

III. To demonstrate the feasibility of central molecular risk stratification of patients with newly diagnosed RMS in the context of a prospective clinical trial.

EXPLORATORY OBJECTIVES:

I. To collect blood and tissue samples for banking at baseline, during treatment, at the end of therapy, and at the time of progression to bank for future research.

II. To describe the methylation array profile of patients with fusion negative, low-risk rhabdomyosarcoma.

III. To describe the outcomes of patients with VLR or LR RMS and MYOD1 or TP53 mutations treated with intensified therapy.

OUTLINE: Patients are assigned to 1 of 2 regimens based on clinical features. Patients with positive mutation status are transitioned to a third regimen, Regimen M.

REGIMEN VA: Patients with VLR RMS receive vincristine intravenously (IV) on day 1 of each cycle and days 8 and 15 of cycles 1, 3, 5, and 7 and dactinomycin IV over 1-5 minutes or over 10-15 minutes on day 1 of each cycle. Treatment repeats every 21 days for 8 cycles in the absence of disease progression or unacceptable toxicity. Patients with MYOD1 or TP53 mutated tumors transition to Regimen M at cycle 2 (if mutation status is determined to be positive at week 3) or cycle 3 (if mutation status is determined to be positive after week 3).

REGIMEN VAC/VA: Patients with LR RMS receive vincristine IV on day 1 of each cycle and days 8 and 15 of cycles 1-3. Patients also receive dactinomycin IV over 1-5 minutes or 10-15 minutes and cyclophosphamide IV over 60 minutes on day 1 of each cycle. Treatment repeats every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive vincristine IV on day 1 of each cycle and days 8 and 15 of cycles 5-7 and dactinomycin IV over 1-5 minutes or over 10-15 minutes on day 1 of each cycle. Treatment repeats every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients with MYOD1 or TP53 mutated tumors transition to Regimen M at cycle 2 (if mutation status is determined to be positive at week 3) or cycle 3 (if mutation status is determined to be positive after week 3). Patients may also undergo radiation therapy at cycle 5.

REGIMEN M: Patients receive vincristine IV on day 1 of each cycle and days 8 and 15 of cycles 2-4, 7-8, and 11-12 and dactinomycin IV over 1-5 minutes or 10-15 minutes on day 1 of cycles 2-5 and 8-14. Patients also receive cyclophosphamide IV over 60 minutes on day 1 of each cycle. Treatment repeats every 21 days for 12-13 cycles in the absence of disease progression or unacceptable toxicity. Patients may also undergo radiation therapy at cycle 5.

Patients undergo computed tomography (CT) scan, magnetic resonance imaging (MRI), bone scan, positron emission tomography (PET) scan and tumor biopsy throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* All patients must be enrolled on APEC14B1 (NCT02402244) and consented to the Molecular Characterization Initiative (Part A) prior to enrollment and treatment on ARST2032 (this trial).
* Patients must be =< 21 years at the time of enrollment.
* Patients must have newly diagnosed embryonal rhabdomyosarcoma (ERMS), spindle cell/sclerosing RMS, or FOXO1 fusion negative alveolar rhabdomyosarcoma (ARMS) (institutional FOXO1 fusion results are acceptable). RMS types included under ERMS include those classified in the 1995 International Classification of Rhabdomyosarcoma (ICR) as ERMS (classic, spindle cell, and botryoid variants), which are reclassified in the 2020 World Health Organization (WHO) classification as ERMS (classic, dense and botryoid variants) and spindle cell/sclerosing RMS (encompassing the historical spindle cell ERMS variant and the newly recognized sclerosing RMS variant). Enrollment in APEC14B1 is required for all patients.

  * All patients will be evaluated for stage and clinical group. Note that clinical group designation assigned at the time of enrollment on study remains unchanged regardless of any second-look operation that may be performed.

    * Patients will be eligible for the very low-risk stratum (Regimen VA) if they have Stage 1, CG I disease.
    * Patients will be eligible for the low-risk stratum (Regimen VAC/VA) if they have Stage 1, CG II disease, Stage 2, CG I or II disease, or Stage 1, CG III (orbit only) disease.
  * Paratesticular Tumors: Staging ipsilateral retroperitoneal lymph node sampling (SIRLNS) is required for all patients >= 10 years of age with paratesticular tumors who do not have gross nodal involvement on imaging.
  * Extremity Tumors: Regional lymph node sampling is required for histologic evaluation in patients with extremity tumors.
  * Clinically or radiographically enlarged nodes must be sampled for histologic evaluation.
* Patients must have a Lansky (for patients =< 16 years of age) or Karnofsky (for patients > 16 years of age) performance status score of >= 50. Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing performance score.
* Peripheral absolute neutrophil count (ANC) >= 750/uL (within 7 days prior to enrollment).
* Platelet count >= 75,000/uL (transfusion independent) (within 7 days prior to enrollment).
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 or a serum creatinine (within 7 days prior to enrollment) based on age/gender as follows:

  * Age: 1 month to < 6 months; Maximum serum creatinine (mg/dL): 0.4 (male) : 0.4 (female)
  * Age: 6 months to < 1 year; Maximum serum creatinine (mg/dL): 0.5 (male) : 0.5 (female)
  * Age: 1 to < 2 years; Maximum serum creatinine (mg/dL): 0.6 (male) : 0.6 (female)
  * Age: 2 to < 6 years; Maximum serum creatinine (mg/dL): 0.8 (male) : 0.8 (female)
  * Age: 6 to < 10 years; Maximum serum creatinine (mg/dL): 1 (male) : 1 (female)
  * Age: 10 to < 13 years; Maximum serum creatinine (mg/dL): 1.2 (male) : 1.2 (female)
  * Age: 13 to < 16 years; Maximum serum creatinine (mg/dL): 1.5 (male) : 1.4 (female)
  * Age >= 16 years; Maximum serum creatinine (mg/dL): 1.7 (male) : 1.4 (female)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) for age (within 7 days prior to enrollment), and

  * If there is evidence of biliary obstruction by the tumor, then the total bilirubin must be < 3 x ULN for age.
  * Note: For the purpose of this study, the ULN for SGPT (ALT) has been set to the value of 45 U/L.
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 135 U/L

  * If there is evidence of biliary obstruction by the tumor, then the total bilirubin must be < 3 x ULN for age
  * Note: For the purpose of this study, the ULN for SGPT (ALT) has been set to the value of 45 U/L
* All patients and/or their parents or legal guardians must sign a written informed consent.
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met.

Exclusion Criteria:

* Patients who have received prior chemotherapy and/or radiation therapy for cancer prior to enrollment. Surgical resection alone of previous cancer(s) is permitted.
* Patients who have received chemotherapy or radiation for non-malignant conditions (e.g., autoimmune diseases) are eligible. Patients must discontinue chemotherapy for non-malignant conditions prior to starting protocol therapy.
* Vincristine is sensitive substrate of the CYP450 3A4 isozyme. Patients must not have received drugs that are moderate to strong CYP3A4 inhibitors and inducers within 7 days prior to study enrollment.
* Patients unable to undergo radiation therapy, if necessary, as specified in the protocol.
* Evidence of uncontrolled infection.
* Female patients who are pregnant since fetal toxicities and teratogenic effects have been noted for several of the study drugs. A pregnancy test is required for female patients of childbearing potential.
* Lactating females who plan to breastfeed their infants.
* Sexually active patients of reproductive potential who have not agreed to use an effective contraceptive method for the duration of their study participation.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 205 (Estimated)
Dates: Start 2022-08-04 (Actual); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Failure free survival (FFS) for very low risk patients | From study enrollment to disease progression, recurrence, or death as a first event, assessed up to 3 years
  The Kaplan-Meier method will be used to estimate 3-year FFS along with 80% log-minus-log transformed confidence limits for very low risk (VLR) patients.
Failure free survival (FFS) for low risk patients | From study enrollment to disease progression, recurrence, or death as a first event, assessed up to 3 years
  The Kaplan-Meier method will be used to estimate 3 year FFS along with 80% log-minus-log transformed confidence limits for low risk (LR) patients.

SECONDARY OUTCOMES:
Overall survival (OS) for very low risk patients | From study entry to death of any cause, assessed up to 5 years
  Log-rank test will be used to compare the OS of patients with VLR rhabdomyosarcoma (RMS) treated with 24 weeks of vincristine, dactinomycin (VA) to the VLR RMS patients from ARST0331 and D9602 with the same inclusion criteria.
Overall survival (OS) for low risk patients | From study entry to death of any cause, assessed up to 5 years
  Log-rank test will be used to compare the OS from LR RMS patients to LR RMS patients from ARST0331 and D9602 with the same inclusion criteria.
Feasibility of central molecular risk stratification of patients assessed by the percentage of patients who have molecular testing results returned by 6 weeks | Up to 24 weeks
  If the percentage of patients who have molecular testing results returned by 6 weeks is >= 80% then the central molecular risk stratification is considered feasible.

OTHER OUTCOMES:
Methylation array profile of patients with fusion negative, low-risk rhabdomyosarcoma | Up to 5 years
  Summary statistics will be used to describe the methylation array profile of patients with fusion negative, low-risk rhabdomyosarcoma. Correlation between methylation patterns and clinical presentation, histology, and genetics will be evaluated.
Descriptive analysis of patients treated on Regimen M | Up to 5 years
  Summary statistics will be used to provide a descriptive analysis of patients treated on Regimen M, including patient demographics, clinical characteristics and outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Josephine H Haduong, Principal Investigator — Children's Oncology Group
Locations (177):
- United States (162):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - USA Health Strada Patient Care Center, Mobile, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - Naval Medical Center -San Diego, San Diego, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Atrium Health Navicent, Macon, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Children's Hospital-Park Ridge, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Northwestern Medicine Central DuPage Hospital, Winfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Wesley Medical Center, Wichita, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Maine Children's Cancer Program, Scarborough, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Corewell Health Children's, Royal Oak, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - UMC Cancer Center / UMC Health System, Lubbock, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Carilion Children's, Roanoke, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (3):
  - Sydney Children's Hospital, Randwick, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Perth Children's Hospital, Perth, Western Australia
- Canada (10):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec
  - CHU de Quebec-Centre Hospitalier de l'Universite Laval (CHUL), Québec
- New Zealand (2):
  - Starship Children's Hospital, Grafton, Auckland
  - Christchurch Hospital, Christchurch